CLINICAL TRIAL: NCT06083831
Title: The Effect of Sequential Feeding for Circadian Rhythm and Gut Flora Rhythm in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Bo Yao,phD, Attending physician, The Affiliated Hospital of Qingdao University
Other Study IDs: QYFYEC2023-108
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Feeding Patterns; Critical Illness; Circadian Rhythm Disorders
MeSH Terms: conditions — Feeding Behavior; Critical Illness; Chronobiology Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sequential feeding group: After achieving ≥80% of the nutrition target calories (25-30 kcal/kg/d) by continuous feeding, continuous feeding was changed into intermittent feeding. The total daily dosage of enteral nutrition was equally distributed during three periods at 7-9:00, 11-13:00 and 17-19:00. The enteral nutritional suspension administered during each period was given at a uniform rate within two hours by an enteral feeding pump. The other times of the day were fasting times.
  Interventions: Other: feeding type
- Continuous feeding group: Patients received continous feeding with a constant velocity by an enteral feeding pump over one day.
  Interventions: Other: feeding type

INTERVENTIONS:
Other: feeding type — In our department, the ICU patients received continuous feeding or sequential feeding. Patients received continuous feeding with a constant velocity by an enteral feeding pump over one day. In sequential feeding type, after achieving ≥80% of the nutrition target calories (25-30 kcal/kg/d), the patients received intermittent feeding. The total daily dosage of enteral nutrition was equally distributed during three periods at 7-9:00, 11-13:00 and 17-19:00. The enteral nutritional suspension administered during each period was given at a uniform rate within two hours by an enteral feeding pump. The other times of the day were fasting times.

SUMMARY:
Circadian rhythms plays an important role for healthy. And critical illness contributes to the disruption of circadian rhythms. Not only right but also feeding can affect the circadian clock gene expression. In a investigators' previous study, some metabolic indicators (the albumin level, total cholesterol level and total bile acid level) and the increases in lymphocyte counts in the sequential feeding group were different from those in the continuous feeding group. Investigators think sequential feeding may adjust circadian clock gene expression for its effect on metabolism and immunity. Moreover, sequential feeding did alter the abundances of some gut microbes to some degree in the investigators' previous study. Investigators think sequential feeding may adjust gut flora rhythms.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly admitted to ICU were eligible for inclusion.

Exclusion Criteria:

* An estimated feeding time of less than 10 days in ICU;
* Diabetes;
* Gastrointestinal disease (gastrointestinal surgery, gastrointestinal bleeding, pancreatitis, Crohn's disease, ulcerative colitis, irritable bowel syndrome);
* Inability to tolerate ≥80% of the nutrition target calories (25-30 kcal/kg/d) with enteral feeding through gastric tube;
* The ability to eat orally at admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
clock genes expression | 7 days feeding
  Genes including BMAL1 CLOCK TIMELESS PER1 and so on
Gut Flora Rhythm | 7 days feeding
  α diversity including shannon index and so on

CONTACTS AND LOCATIONS:
Overall Officials: bo yao, Dr., Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The affiliated hospital of qingdao university, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided